CLINICAL TRIAL: NCT02870361
Title: Einfluss Der zentralnervösen Insulinsensitivität Auf Die Insulinsekretion
Brief Title: Influence of Central Nervous Insulin Sensitivity on Insulin Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 086/2016BO1
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Insulin Secretion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin nasal spray (Active Comparator): 160 Units of human insulin as nasal spray
  Interventions: Drug: intranasal insulin
- Placebo nasal spray (Placebo Comparator): Nasal spray containing placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intranasal insulin
  Arms: Insulin nasal spray
Drug: Placebo
  Arms: Placebo nasal spray

SUMMARY:
Insulin resistance is a central pathophysiological component of type 2 diabetes and is associated with a high risk of cardiovascular disease. The tissue in which it manifests are mainly muscle, liver, and adipose tissue. Since the transport of glucose to the brain is independent of insulin, this organ has traditionally not been studied in this regard. In animal experiments, however, knockout of the insulin receptor in the brain leads to obesity and peripheral insulin resistance. This finding of insulin action in the brain could also be confirmed in human studies.

The investigators intend to investigate whether central nervous insulin action affects insulin secretion in humans. For this purpose, nasal insulin and placebo are administered 15 minutes before a hyperglycemic hyperinsulinemic clamps, which stimulate insulin secretion. Insulin sensitivity of the brain is measured by a an established protocol with functional magnetic resonance imaging before and after nasal insulin administration.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≤6.0%
* normal glucose tolerance during 75g oral glucose tolerance test (OGTT)

Exclusion Criteria:

* Not removable metal parts in or on the body
* manifest cardiovascular disease
* claustrophobia
* recent surgery (less than 3 months)
* Simultaneous participation in other studies
* Acute disease or infection within the last 4 weeks
* neurological and psychiatric disorders
* treatment with centrally acting drugs
* hemoglobin Hb <13g / dl
* Hypersensitivity to any of the substances used

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Insulin secretion assessed as serum C-peptide levels during a hyperglycemic clamp | 0-10 min during hyperglycemic clamp and 10-90 min during hyperglycemic clamp

SECONDARY OUTCOMES:
Correlation with brain insulin sensitivity | 15-30 minutes post insulin nasal spray
  Correlation of regional brain insulin sensitivity with the change of pancreatic insulin secretion due to central action of insulin. Changes in regional cerebral blood flow from before to after intranasal insulin administration will be assessed by functional magnetresonance imaging (fMRI)
Differential effects in lean and overweight | 0-10 min during hyperglycemic clamp and 10-90 min during hyperglycemic clamp
  Differences in the effect of nasal insulin versus placebo on C-peptide levels during a hyperglycemic clamp between lean and overweight men will be assessed.
Correlation with autonomous nervous system activity | 10 - 150 minutes post nasal spray
  Correlation of the change in pancreatic insulin secretion by central insulin action with the simultaneous change of the autonomous nervous system (measured by heart rate variability).
Peripheral insulin sensitivity | 10-90 min and 70-90 min during hyperglycemic clamp
  Effect of nasal insulin versus placebo on peripheral insulin sensitivity assessed by hyperglycemic hyperinsulinemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heni M, Wagner R, Willmann C, Jaghutriz BA, Vosseler A, Kubler C, Hund V, Scheffler K, Peter A, Haring HU, Preissl H, Kullmann S, Fritsche A. Insulin Action in the Hypothalamus Increases Second-Phase Insulin Secretion in Humans. Neuroendocrinology. 2020;110(11-12):929-937. doi: 10.1159/000504551. Epub 2019 Nov 5. PMID 31689708